CLINICAL TRIAL: NCT00636051
Title: Evidence-Based Practice (EBP) Awareness Project: Peer-to-Peer Dissemination
Status: Completed | Type: Observational
Sponsor: State University of New York - Upstate Medical University (Other)
Responsible Party: Priscilla Sandford Worral, Coordinator of Nursing Research, University Hospital, SUNY Upstate Medical University
Other Study IDs: #5166
Record Dates: First submitted 2008-03-07; First posted 2008-03-14 (Estimated); Last update posted 2009-06-09 (Estimated); Status verified 2009-06

CONDITIONS: Evidence-Based Medicine
Keywords: evidence based practice beliefs; evidence based practice implementation; evidence based practice dissemination

STUDY DESIGN:
Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- 1: staff Registered Nurses receiving EBP peer mentoring
- 2: staff Registered Nurses not receiving EBP peer mentoring

SUMMARY:
The purpose of this study is to evaluate the effectiveness of the introduction of an EBP text for Nursing Research Council (NRC) members to use with RN staff to increase staff belief in, knowledge of and implementation of EBP in providing patient care. The theory that will drive this study is Disciplined Clinical Inquiry (DCI).

The current study will use a quasi-experimental design plus DCI to engage unit RN staff in deciding how they might learn about EBP in a feasible, useful way. After collection of baseline data, the NRC member will introduce the text + solicit staff input into a plan for using the text to increase understanding of EBP and use of evidence to make practice changes on her/his own unit. Another unit in that service line or under the same Service Line Administrator will serve as a comparison unit. Data collection will be conducted again after 4 and 12 weeks. At the 12 week point, the NRC member will introduce the text + solicit staff input for a plan on the comparison unit. Data collection will be conducted on the comparison unit at 16 weeks, and again on both units at 24 weeks. At the 24 week point, additional units will be added and the process repeated until all units represented on the NRC have been included.

Outcome measures will include: EBP belief and EBP implementation scales (Melnyk & Fineout-Overholt, 2003); EBP knowledge cognitive test; # of lit searches conducted by unit RN staff ; # of requests for library support for lit searches or to obtain search-related articles: # of unit clinical policies with documented levels of evidence & research references. EBP belief, EBP implementation and EBP knowledge variables will be analyzed at both individual and unit levels of analysis. All other variables will be measured at the unit level of analysis. Additional unit level variables will include the following data collected annually as part of the National Database for Nursing Quality Indicator (NDNQI) RN satisfaction survey: satisfaction with RN-RN interaction, satisfaction with autonomy, satisfaction with practice decision-making, perceived quality of care delivered on the unit.

The primary statistical procedures for analysis will be ANCOVA, ANOVAwith repeated measures, and logistic regression.

ELIGIBILITY:
Inclusion Criteria:

* over 18 yrs of age
* employed by Upstate
* full or parttime on unit represented on Nursing Research Council

Exclusion Criteria:

* employed by an agency other than Upstate
* working on a unit not represented on the Nursing Research Council

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: All RN staff & RN patient service leaders (PSLs) who are over 18 years of age, employed by Upstate and working full or parttime on direct care units within service lines represented on the Nursing Research Council (NRC) will be invited to participate. This target population includes approximately 551 staff RNs & PSLs. We expect to enroll a minimum of 5 and as many as 15 RNs on the 29 nursing units over the course of the study for a sample size between 145 and 435
Sampling Method: Probability Sample
Enrollment: 91 (Actual)
Dates: Start 2005-02; Primary Completion 2006-11 (Actual); Study Completion 2006-11 (Actual)

PRIMARY OUTCOMES:
EBP Beliefs | baseline, 4 wks, 8 wks, 12 wks, 24 wks

SECONDARY OUTCOMES:
EBP Implementation | baseline, 4 wks, 8 wks, 12 wks, 24 wks,

CONTACTS AND LOCATIONS:
Overall Officials: Priscilla S Worral, PhD, RN, Principal Investigator — State University of New York - Upstate Medical University